CLINICAL TRIAL: NCT05705557
Title: Assessment of Efficacy of ABSOLOK™ Clip System-RFP-2021-01 in Achieving BIliostasis During Parenchymal Transection for Open Liver Resection
Brief Title: Efficacy of ABSOLOK™ Clip System-RFP-2021-01 in Open Liver Resection
Acronym: EBILROK
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 5139
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bile Leak
Keywords: Liver resection; Hepatectomy; Absolok; Bile Leak; Laparotomy; Open Liver resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OPEN Liver Resection: Patients undergoing laparotomic (OPEN) Liver Resection
  Interventions: Device: ABSOLOK™ Clip System

INTERVENTIONS:
Device: ABSOLOK™ Clip System — Use of ABSOLOK™ Clip System during parenchymal transection for open liver resection

SUMMARY:
The purpose of this prospective observational study is to evaluate the incidence of Post-Operative Bile Leakage (POBL) using the ABSOLOK™ Clip System during liver parenchymal resection by evaluating the intraoperative and short-term postoperative results. In addition, it will attempt to determine the factors that determine the surgeon's peripheral glissonian pedicle closure method and economic outcomes.

DETAILED DESCRIPTION:
Over the last two decades, significant advances have been made in hepatectomy because of advancements in surgical techniques and improvement on parenchymal transection. Modern liver surgeon must be equipped with excellent theoretical and clinical skills to perform a safe liver resection. Despite significant technical advancements in the field of liver surgery, bile leakage remains a significant postoperative morbidity. Although the exact post-hepatectomy bile leakage site is not clear, bile leakage reportedly occurs in 3-12% according to the kind of resection.

Recently, in a large multicenter retrospective series, including 13.379 resected patients, the overall incidence of post-operative bile leakage (POBL) is 6%, significantly higher after open versus laparoscopic approach, respectively 9,4% vs 3,1% (p<0.001). POBL was defined according to the 2010 International Study Group of Liver Surgery (ISGLS) and it was categorized in three grades of severity (grade A, B, C) and clinically relevant POBL (CR-POBL) was defined as grade B and C. CR-POBL is associated with increased length of post-operative stay and can be associated with subsequent severe complications such as intra-abdominal abscess, peritonitis, and sepsis. In the case of anatomical liver resection, most of the leakage points are observed around the hilar Glissonean stump and not at the peripheral parenchymal cutting plane, because parenchymal resection is usually performed along the intersegmental plane.

Recently, parenchyma-sparing hepatectomy (PSH) has become a gold standard treatment for colorectal liver metastases (CLM). PSH is associated with better perioperative outcomes without compromising oncological outcomes and given the relatively high incidence of hepatic parenchymal recurrence, the PSH treatment offers a greater opportunity of repeat resection for intrahepatic recurrences.

Anatomic resection (AR) remains the gold standard surgical treatment for hepatocellular carcinoma (HCC) in patients with a well-preserved liver function because postoperative recurrence is usually caused by micrometastases around the tumor therefore resecting the tumor-bearing portal branches and the corresponding liver parenchyma achieving better local control. US-guided limited resection (LR) and AR may be chosen and/or combined by the surgeon for the other surgical indications. Most of the leakage points are observed at the peripheral parenchymal cutting plane despite the liver parenchymal transection was carried out using the ultrasonic dissector and all peripheral glissonian pedicles (≥ 2-3 mm) were separately isolated, clipped or ligated and transected.

The aim of the prospective study is to assess the incidence of POBL using ABSOLOK™ Clip System during parenchymal liver transection, evaluating intra-operative and short-term post-operative results. In addition, the factors that determine the surgeon's peripheral glissonian pedicle closure method and cost results will be tried to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Subject has given his informed consent and signed consent;
* Patients undergoing open liver resection.

Exclusion Criteria:

* Surgery made in emergency;
* Surgery by laparoscopy;
* Need to perform a bilio-digestive anastomosis;
* Preoperative jaundice (total bilirubin > 3 mg/mL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparotomic (open) liver resection or re-resection for any underlying disease. The list of underlying diseases is the following (but might not be limited to):
  * Colorectal liver metastases;
  * Liver metastases from other primary malignancy (Breast, Ovarian, Neuroendocrine Tumors, Adrenal, Non-neuroendocrine Tumors, Other);
  * Intrahepatic Cholangiocarcinoma;
  * Gallbladder Cancer;
  * Hepatocellular Carcinoma;
  * Benign Tumors (Hepatic Adenoma, Haemangioma, Focal nodular hyperplasia);
  * Intrahepatic Bile Duct dilation and/or intrahepatic lithiasis;
  * Hidatid Cyst.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Overall Post-Operative Bile Leakage (POBL) using ABSOLOK™ Clips during liver resection | 90 days
  Participants will be followed for the duration of hospital stay and Follow Up

SECONDARY OUTCOMES:
Duration of POBL (Post-operative bile leakage) and the timing of drainage removal | 90 days
  Participants will be followed for the duration of hospital stay and Follow Up
Additional maneuvers for treat biliary fistula | 90 days
  Participants will be followed for the duration of hospital stay and Follow Up
Lenght of post-operative stay | 90 days
  Participants will be followed for the duration of hospital stay
Rate of post-operative Morbidity | 90 days
  Participants will be followed for the duration of hospital stay and Follow Up
Rate of post-operative Mortality | 90 days
  Assessment of mortality during the hospitalization or Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Felice Giulante, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torzilli G, McCormack L, Pawlik T. Parenchyma-sparing liver resections. Int J Surg. 2020 Oct;82S:192-197. doi: 10.1016/j.ijsu.2020.04.047. Epub 2020 Apr 23. PMID 32335245
- [Background] Martin AN, Narayanan S, Turrentine FE, Bauer TW, Adams RB, Stukenborg GJ, Zaydfudim VM. Clinical Factors and Postoperative Impact of Bile Leak After Liver Resection. J Gastrointest Surg. 2018 Apr;22(4):661-667. doi: 10.1007/s11605-017-3650-4. Epub 2017 Dec 15. PMID 29247421
- [Background] Brooke-Smith M, Figueras J, Ullah S, Rees M, Vauthey JN, Hugh TJ, Garden OJ, Fan ST, Crawford M, Makuuchi M, Yokoyama Y, Buchler M, Weitz J, Padbury R. Prospective evaluation of the International Study Group for Liver Surgery definition of bile leak after a liver resection and the role of routine operative drainage: an international multicentre study. HPB (Oxford). 2015 Jan;17(1):46-51. doi: 10.1111/hpb.12322. Epub 2014 Jul 24. PMID 25059275
- [Background] Gorgec B, Cacciaguerra AB, Aldrighetti LA, Ferrero A, Cillo U, Edwin B, Vivarelli M, Lopez-Ben S, Besselink MG, Abu Hilal M; International Study Group of Bile Leakage after Liver Surgery. Incidence and Clinical Impact of Bile Leakage after Laparoscopic and Open Liver Resection: An International Multicenter Propensity Score-Matched Study of 13,379 Patients. J Am Coll Surg. 2022 Feb 1;234(2):99-112. doi: 10.1097/XCS.0000000000000039. PMID 35213428
- [Background] Koch M, Garden OJ, Padbury R, Rahbari NN, Adam R, Capussotti L, Fan ST, Yokoyama Y, Crawford M, Makuuchi M, Christophi C, Banting S, Brooke-Smith M, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Nimura Y, Figueras J, DeMatteo RP, Buchler MW, Weitz J. Bile leakage after hepatobiliary and pancreatic surgery: a definition and grading of severity by the International Study Group of Liver Surgery. Surgery. 2011 May;149(5):680-8. doi: 10.1016/j.surg.2010.12.002. Epub 2011 Feb 12. PMID 21316725
- [Background] Deng G, Li H, Jia GQ, Fang D, Tang YY, Xie J, Chen KF, Chen ZY. Parenchymal-sparing versus extended hepatectomy for colorectal liver metastases: A systematic review and meta-analysis. Cancer Med. 2019 Oct;8(14):6165-6175. doi: 10.1002/cam4.2515. Epub 2019 Aug 28. PMID 31464101
- [Background] Sun Z, Li Z, Shi XL, He XW, Chen J, Song JH. Anatomic versus non-anatomic resection of hepatocellular carcinoma with microvascular invasion: A systematic review and meta-analysis. Asian J Surg. 2021 Sep;44(9):1143-1150. doi: 10.1016/j.asjsur.2021.02.023. Epub 2021 Mar 23. PMID 33766529
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Mohkam K, Farges O, Vibert E, Soubrane O, Adam R, Pruvot FR, Regimbeau JM, Adham M, Boleslawski E, Mabrut JY; Association de Chirurgie Hepato-Biliaire et de Transplantation (ACHBT) French Hepatectomy Study Group. Risk score to predict biliary leakage after elective liver resection. Br J Surg. 2018 Jan;105(1):128-139. doi: 10.1002/bjs.10647. Epub 2017 Nov 13. PMID 29131313
- [Background] Maulat C, Regimbeau JM, Buc E, Boleslawski E, Belghiti J, Hardwigsen J, Vibert E, Delpero JR, Tournay E, Arnaud C, Suc B, Pessaux P, Muscari F. Prevention of biliary fistula after partial hepatectomy by transcystic biliary drainage: randomized clinical trial. Br J Surg. 2020 Jun;107(7):824-831. doi: 10.1002/bjs.11405. Epub 2020 Jan 9. PMID 31916605
- [Background] Vigano L, Torzilli G, Troisi R, Aldrighetti L, Ferrero A, Majno P, Toso C, Figueras J, Cherqui D, Adam R, Kokudo N, Hasegawa K, Guglielmi A, Krawczyk M, Giuliante F, Hilal MA, Costa-Maia J, Pinna AD, Cescon M, De Santibanes E, Urbani L, Pawlik T, Costa G, Zugna D; CLISCO group. Minor Hepatectomies: Focusing a Blurred Picture: Analysis of the Outcome of 4471 Open Resections in Patients Without Cirrhosis. Ann Surg. 2019 Nov;270(5):842-851. doi: 10.1097/SLA.0000000000003493. PMID 31569127
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660